CLINICAL TRIAL: NCT01920282
Title: Effect of Nebivolol and Lifestyle Modification on Large Artery Stiffness in Middle-Aged and Older Hypertensive Adults
Brief Title: Nebivolol, Lifestyle Modification and Arterial Stiffness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Kevin Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: nebstiff
Record Dates: First submitted 2013-07-18; First posted 2013-08-09 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Nebivolol (Active Comparator): Subjects will be provided with daily 5 mg of nebivolol for the first 2 weeks. Subjects receive additional daily doses of 10 mg nebivolol for the remainder of the study period. The dose remains at 5 mg per day, however, if BP falls below 110/70 during the first 2 weeks. Subjects will continue taking the drug during the 2-week follow-up period.
  Interventions: Drug: Nebivolol
- Lifestyle Modification (Active Comparator): Subjects will receive weekly lifestyle counseling by a registered dietitian to ensure adequate progress and compliance. Sample menus, 14-days of meal plans, and grocery shopping lists are provided to each individual. Individuals were instructed to reduce their daily caloric intake by 500-1000 calories and to perform a minimum of 150 minutes per week of moderate-intensity physical activity or 3000 steps/day above baseline levels. The diet plan conformed to the Dietary Approach to Stop Hypertension dietary guidelines emphasizing low fat dairy products, fruits and vegetable and contained 55% calories as carbohydrates, 30% calories as fat, and 15% calories as protein. Sodium consumption was set at 2,400 mg/day for all subjects.
  Interventions: Other: Lifestyle Modification
- Nebivolol plus Lifestyle Modification (Experimental): Subjects begin with 5 mg/day of nebivolol and increase to 10 mg/day if brachial blood pressure is greater than 120/80 mmHg during the first 2 weeks of therapy. Subjects also receive weekly lifestyle counseling by a registered dietitian to ensure adequate progress and compliance. Sample menus, 14-days of meal plans, and grocery shopping lists are provided to each individual. Individuals will be instructed to reduce their daily caloric intake by 500-1000 calories and to perform a minimum of 150 min/wk of moderate-intensity physical activity or 3000 steps/day above baseline levels. The diet plan conforms to the Dietary Approaches to Stop Hypertension dietary guidelines emphasizing low fat dairy products, fruits and vegetable and contains 55% calories as carbohydrates, 30% calories as fat, and 15% calories as protein with sodium consumption set at 2,400 mg/day for all subjects.
  Interventions: Other: Nebivolol plus Lifestyle Modification

INTERVENTIONS:
Drug: Nebivolol
  Other Names: Bystolic
  Arms: Nebivolol
Other: Lifestyle Modification
  Other Names: Weight loss; Sodium restriction; Physical activity
  Arms: Lifestyle Modification
Other: Nebivolol plus Lifestyle Modification
  Other Names: Bsytolic; Weight Loss; Sodium restriction; Physical activity
  Arms: Nebivolol plus Lifestyle Modification

SUMMARY:
Numerous anti-hypertensive drugs have been reported to be efficacious in reducing central arterial stiffness and these effects may contribute to improved outcomes in hypertensive patients. However, the results of several studies suggest that beta-blockers may actually increase arterial stiffness. In contrast, there is limited evidence to suggest that nebivolol, a third generation beta-blocker that augments release of vascular nitric oxide, reduces central arterial stiffness in hypertensive individuals. Unfortunately, only a few studies have addressed this issue and all of these studies relied on indirect, blood pressure dependent measures of arterial stiffness. In addition, none of these studies focused on middle-aged and older, obese hypertensives, a population with accelerated arterial stiffening and at risk for cardiovascular diseases. Thus, the potential utility of nebivolol as a therapy to reduce large artery stiffness, particularly among the latter population, remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 hypertension
* 40-75 years
* Weight stable (+/-2 kg)
* Sedentary to recreationally active
* Willing to be randomized to one of three arms
* Verbal and written consent
* Approval by medical director

Exclusion Criteria:

* Blood pressure outside stated range
* Diabetes or taking diabetes medications
* Total cholesterol >6.2 mmol/L; triglycerides >4.5 mmol/L
* Past or current ischemic heart disease, stroke, respiratory disease, endocrine or metabolic disease, neurological disease, or hematological-oncological disease
* Medications (including but not limited to antihypertensives, statins or other with anti-inflammatory actions) or antioxidant vitamins or supplements
* Known allergy or hypersensitivity to nebivolol or any of its components
* Inability to perform regular physical activity or participate in other components of lifestyle modification
* Pregnant or planning to become pregnant

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Davy, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University

RESULTS

PARTICIPANT FLOW:
Groups:
- Nebivolol: Subjects will be provided with daily 5 mg of nebivolol for the first 2 weeks. Subjects receive additional daily doses of 10 mg nebivolol for the remainder of the study period. The dose remains at 5 mg per day, however, if BP falls below 110/70 during the first 2 weeks. Subjects will continue taking the drug during the 2-week follow-up period.
  Nebivolol
- Lifestyle Modification: Subjects will receive weekly lifestyle counseling by a registered dietitian to ensure adequate progress and compliance. Sample menus, 14-days of meal plans, and grocery shopping lists were provided to each individual. Individuals were instructed to reduce their daily caloric intake by 500-1000 calories and to perform a minimum of 150 minutes per week of moderate-intensity physical activity or 3000 steps/day above baseline levels. The diet plan conformed to the Dietary Approach to Stop Hypertension dietary guidelines emphasizing low fat dairy products, fruits and vegetable and contained 55% calories as carbohydrates, 30% calories as fat, and 15% calories as protein21. Sodium consumption was set at 2,400 mg/day for all subjects.
  Lifestyle Modification
- Nebivolol Plus Lifestyle Modification: Subjects began with 5 mg/day of nebivolol and increased to 10 mg/day if brachial blood pressure was greater than 120/80 mmHg during the first two weeks of therapy. Subjects also received weekly lifestyle counseling by a registered dietitian to ensure adequate progress and compliance. Sample menus, 14-days of meal plans, and grocery shopping lists were provided to each individual. Individuals were instructed to reduce their daily caloric intake by 500-1000 calories and to perform a minimum of 150 minutes per week of moderate-intensity physical activity or 3000 steps/day above baseline levels. The diet plan conformed to the Dietary Approaches to Stop Hypertension dietary guidelines emphasizing low fat dairy products, fruits and vegetable and contained 55% calories as carbohydrates, 30% calories as fat, and 15% calories as protein21. Sodium consumption was set at 2,400 mg/day for all subjects.
  Nebivolol plus Lifestyle Modification
Period: Overall Study
Arm/Group | Nebivolol | Lifestyle Modification | Nebivolol Plus Lifestyle Modification
Started | 15 | 15 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Lifestyle Modification | Nebivolol Plus Lifestyle Modification | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: yr] | 57.7 (3.1) | 52.7 (2.2) | 58.4 (2.2) | 56.3 (2.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 12 | 36
  >=65 years | 1 | 5 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 23
  Male | 8 | 7 | 7 | 22
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 45
Supine blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 146 (1.4) | 138 (3.1) | 142 (2.6) | 142 (2.37)
Supine heart rate (bpm) [Mean (Standard Deviation); unit: bpm] | 64 (1) | 67 (3) | 66 (2) | 66 (2)

OUTCOME MEASURES:

1. Primary Outcome: Beta-stiffness Index
Description: Longitudinal B-mode images of the left common carotid artery diameter (1-2 cm proximal to the carotid bulb) were obtained over 15 consecutive cardiac cycles. Brachial blood pressure was measured via an automated sphygmomanometer. Quantification of systolic and diastolic carotid artery diameters were analyzed with the Vascular Research Tools 5 software program. Beta-stiffness index was calculated as: Beta = ln(P1/P0)/((D1-D0)/D0), where D0 represents the minimal diameter recorded during diastole, D1 represents the maximal diameter recorded during systole, P0 represents the pressure measured during diastole, and P1 represents the pressure measured during systole.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Nebivolol | Lifestyle Modification | Nebivolol Plus Lifestyle Modification
Number analyzed (Participants) | 15 | 15 | 15
Arbitrary units | -2.03 (0.6) | -1.87 (0.83) | -2.51 (0.9)

2. Secondary Outcome: Insulin Sensitivity (HOMA-IR)
Description: The HOMA index was calculated as the product of plasma blood glucose and insulin divided by 22.5.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Nebivolol | Lifestyle Modification | Nebivolol Plus Lifestyle Modification
Number analyzed (Participants) | 15 | 15 | 15
Arbitrary units | -0.36 (0.33) | -1.98 (1.43) | -2.12 (0.73)

3. Other Pre Specified Outcome: Oxidized LDL Concentration
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nebivolol | Lifestyle Modification | Nebivolol Plus Lifestyle Modification
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No